CLINICAL TRIAL: NCT00077948
Title: A Phase III, Randomized, Double-Blind, Double Placebo-Controlled, Multicenter, Three Parallel Group Study of Enoximone Plus Extended-Release Metoprolol Succinate in Advanced CHF Subjects Previously Intolerant to Beta-Blocker Treatment
Brief Title: Enoximone Plus Extended-Release Metoprolol Succinate in Subjects With Advanced Chronic Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMPOWER (Protocol My-023)
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure, Congestive
Keywords: positive inotrope; enoximone; beta-blocker; intolerant
MeSH Terms: conditions — Heart Failure | interventions — Enoximone; Metoprolol

ARMS (3):
- active enoximone plus active ER metoprolol (Experimental)
  Interventions: Drug: Enoximone; Drug: Metoprolol succinate
- placebo enoximone plus active ER metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol succinate; Drug: Placebo to match enoximone
- placebo enoximone plus placebo ER metoprolol (Placebo Comparator)
  Interventions: Drug: Placebo to match enoximone; Drug: Placebo to match metoprolol succinate

INTERVENTIONS:
Drug: Enoximone — Enoximone administered orally
  Arms: active enoximone plus active ER metoprolol
Drug: Metoprolol succinate — Metoprolol succinate administered orally
  Arms: active enoximone plus active ER metoprolol; placebo enoximone plus active ER metoprolol
Drug: Placebo to match enoximone — Placebo to match match enoximone administered orally
  Arms: placebo enoximone plus active ER metoprolol; placebo enoximone plus placebo ER metoprolol
Drug: Placebo to match metoprolol succinate — Placebo to match metoprolol succinate administered orally
  Arms: placebo enoximone plus placebo ER metoprolol

SUMMARY:
Beta-blocker medications have been shown to improve heart function and prolong the lives of patients with chronic heart failure (CHF). Some people with advanced CHF have difficulty taking beta-blocker medications due to troublesome side effects, such as low blood pressure and/or low heart rate, severe tiredness, dizziness, or shortness of breath. In other words, they have difficulty tolerating beta-blocker medications. The purpose of this study is to determine if enoximone can improve a patient's ability to tolerate a beta-blocker medication.

DETAILED DESCRIPTION:
Over the last decade, it has become evident that certain beta-blocking agents (beta-blockers) exert a favorable effect on the natural history of mild to moderate chronic heart failure (CHF), including reducing mortality and hospitalization rate. However, as heart failure becomes more severe, beta-blockers become difficult to administer because of myocardial depression leading to hemodynamic intolerance. A recent clinical study demonstrated that subjects who could not tolerate the beta-blocker metoprolol experienced improved tolerability when low-dose, oral enoximone was administered prior to the introduction of metoprolol and during ongoing treatment. This study will investigate the hypotheses that by stabilizing subjects on enoximone first, advanced CHF subjects who are intolerant of beta-blockade will be able to 1) tolerate the effects of beta-blocker therapy, and 2) have clinical benefit that is due to the combination of both enoximone and extended-release metoprolol succinate (ER metoprolol). Support for these hypotheses will be sought by demonstrating that, as compared to placebo, low-dose, oral enoximone plus ER metoprolol will increase left ventricular ejection fraction (LVEF), improve symptoms of heart failure, and improve submaximal exercise tolerance in subjects with CHF.

ELIGIBILITY:
Inclusion criteria

In order to be considered an eligible subject, all of the following entry criteria must be met:

* Subjects must be competent to provide informed written consent. Subjects must sign an IRB/IEC approved informed consent form prior to the initiation of any study procedures.
* Subjects must be 18 years of age or older.
* Subjects must have ischemic or nonischemic cardiomyopathy with symptoms of NYHA Class III or IV chronic heart failure.
* Subjects must have a LVEF of less than or equal to 35%, measured within 60 days of the Screening Visit. LVEF must be assessed by radionuclide ventriculography (MUGA). If the subject has experienced any cardiovascular events, has undergone any interventions, or received any changes in treatment that may have affected LV function since the most recent EF measurement, an LVEF measurement must be completed prior to the subject being randomized.
* Subjects must have a left ventricular end diastolic dimension (LVEDD) of >2.7 cm/m2 as measured by 2-D ECHO within 12 months of the Screening Visit.
* Subjects must be on optimal conventional heart failure therapy (with the exception of a beta-blocker), including an ACEI for at least 30 days prior to the Screening Visit, or the subject must have had a trial of an ACEI and proven to be intolerant, or the subject must be taking an ARB for at least 30 days prior to the Screening Visit or proved to be intolerant. Optimal conventional therapy may also include spironolactone, digitalis glycosides, diuretics, or other vasodilators.
* Subjects must have failed the initiation, or the up-titration, of a beta-blocker drug due to hemodynamic intolerance within 12 months prior to the Screening Visit. Failure to tolerate beta-blockade for hemodynamic reasons is defined as worsening signs and symptoms of chronic heart failure, hypotension accompanied with symptoms, or evidence of organ hypoperfusion, which in the judgment of the treating physician precluded further treatment with the beta-blocker. This beta-blocker intolerance must have been documented prior to Screening, and a narrative description of the intolerance must be approved by Myogen prior to Randomization.

Exclusion criteria

Subjects who meet any one of the following criteria will be deemed ineligible for participation in the study:

* Subjects with CHF due to or associated with uncorrected primary valvular disease, uncorrected thyroid disease, obstructive/hypertrophic cardiomyopathy, pericardial disease, amyloidosis, active myocarditis, malfunctioning artificial heart valve, uncorrected congenital heart disease, isolated right-sided heart failure, or primary pulmonary hypertension.
* Subjects who have undergone a cardiac revascularization, valvular surgery, or bi-ventricular resynchronization procedure within 60 days prior to the Screening Visit.
* Subjects listed for heart transplantation who are expected to be transplanted within 6 months of randomization.
* Subjects who have had a myocardial infarction within 90 days prior to the Screening Visit.
* Subjects with an ECG recorded at the Screening Visit showing any of the following: 1) evidence of transmural ischemia (dynamic ST elevation or ST elevation associated with ischemic symptoms), or 2) ventricular tachycardia (VT) or premature ventricular complexes (PVCs) associated with symptoms, or 3) VT of greater than or equal to 6 beats
* Subjects with sustained (>15 seconds) VT, unless precipitated by an event such as an acute myocardial infarction, induction by catheter placement, or by an electrophysiology procedure, or addressed by AICD placement.
* Subjects with an AICD that has fired for any ventricular arrhythmia within 90 days of the Randomization Visit.
* Subjects with a documented diagnosis of angina that meets either of the following criteria: 1) angina diagnosed as unstable at any time within the 60 days prior to the Screening Visit or 2) angina is the primary symptom that limits daily physical activity
* Subjects who have had ventricular reduction surgery or cardiac myoplasty.
* Subjects on a mechanical assist device.
* Subjects with evidence of a concomitant disease that may interfere with the natural course of the subject's underlying heart failure for the duration of the trial.
* Subjects having a concomitant life-threatening disease for which their life expectancy is estimated to be less than one year.
* Subjects with uncontrolled insulin-dependent diabetes mellitus with a history of frequent hypoglycemic episodes or frequent hospitalizations for hyperglycemia.
* Subjects on the following concomitant medications at the time of Screening are excluded from participating in the study: 1) Calcium antagonists other than amlodipine or felodipine; 2) Flecainide, encainide, propafenone, sotalol, dofetilide or disopyramide; 3) Subjects receiving i.v. positive inotropic agents within seven days of the Screening Visit or Randomization Visit; 4) Subjects receiving a human BNP, including nesiritide, within seven days of the Screening Visit or Randomization Visit; 5) Subjects receiving oral or i.v. type-III PDE inhibitors within seven days of the Screening Visit or Randomization Visit.
* Subjects with a contraindication to treatment with a positive inotropic agent (defined as a serious adverse event attributed to previous treatment with a positive inotrope).
* Subjects with a known contraindication to beta-blocker therapy. This may include beta-agonist-dependent chronic obstructive pulmonary disease or asthma, a heart rate <55 BPM, the presence of second- or third-degree heart block without an implanted pacemaker, and first-degree heart block with a PR interval >220 milliseconds.
* Subjects with active hepatic (screening serum total bilirubin greater than or equal to 3.0 mg/dL), renal (screening serum creatinine greater than or equal to 2.0 mg/dL), hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease, which in the opinion of the Investigator, may adversely affect the safety and efficacy of the study drug or the life span of the subject.
* Subjects known to abuse or actively abusing alcohol or illicit drugs. Abuse of alcohol is defined as the usual daily intake of more than 100 grams of ethanol per day, or more than approximately 6 twelve-ounce bottles of beer, one 750 mL bottle of wine or 250 mL of 80 proof spirits.
* Subjects with a serum potassium <4.0 mEq/L or >5.5 mEq/L at Screening.
* Subjects with a serum digoxin of >1.2 ng/mL at Screening are excluded.
* Pregnant women and women at risk of becoming pregnant (i.e., not using effective methods of birth control).
* Subjects who have participated in a clinical trial involving another investigational drug or device within 30 days of the Screening Visit or at any time during the study.
* Subjects who have demonstrated noncompliance with previous medical regimens.
* Subjects who are hospitalized at the time of the Randomization Visit and are not hemodynamically stable, or for whom there is an acute cardiac or non-cardiac illness that requires further hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 2003-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants experiencing improved metoprolol tolerability when coadministered with enoximone | Baseline to Week 36
  Improved tolerability measured by increased left ventricular ejection fraction (LVEF), improvement of heart failure symptoms, and improvement in submaximal exercise tolerance.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - University of Utah, Salt Lake City, Utah